CLINICAL TRIAL: NCT07274943
Title: Patterns Of End-To-Side Arterial Suturing To The Iliac Arteries In Living Donor Kidney Transplantation
Brief Title: End-to-Side Interrupted Versus Continuous Arterial Suturing in Living Donor Kidney Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aly Adel Abdelhamid Ahmed Elyounsy, Resident at the Department of Urology, Assiut University, Assiut University
Other Study IDs: Arterial suturing in kidney
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Suture Techniques; Suture, Interrupted; Continuous Suture; Kidney Transplant
Keywords: donor kidney transplantation; end-to-side arterial suturing; iliac arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Interrupted Arterial Suturing: Adult living donor kidney transplant recipients whose renal artery is anastomosed end-to-side to the external or common iliac artery using interrupted 6/0 Prolene sutures as part of standard surgical practice.
- Continuous Arterial Suturing: Adult living donor kidney transplant recipients whose renal artery is anastomosed end-to-side to the external or common iliac artery using continuous 6/0 Prolene sutures as part of standard surgical practice.

SUMMARY:
This study will compare two standard ways of stitching the kidney artery to the iliac artery in adults receiving a living donor kidney transplant. The two techniques are interrupted suturing and continuous suturing. The study will review past transplant cases and follow new patients at Assiut University Urology Hospital. For each patient, the team will record details of the operation, blood flow in the kidney artery, kidney function, and any surgical or vascular complications during the first three months after surgery. The main goals are to see whether one suturing pattern shortens cold ischemia time and improves early blood flow measurements, and to explore how these techniques affect early graft function, complication rates, and short-term graft and patient survival.

DETAILED DESCRIPTION:
This observational study evaluates whether different patterns of arterial suturing during kidney transplantation influence short-term graft function and vascular outcomes in adult living donor kidney recipients. The study compares interrupted versus continuous end-to-side arterial anastomosis to the iliac arteries using standardized surgical and postoperative care pathways.

The research is designed as a combined retrospective and prospective non-randomized comparative cohort study conducted at the Assiut Kidney Transplantation Unit, Assiut University Urology Hospital. Adult patients who underwent or will undergo living donor kidney transplantation from November 2015 onward are assigned to one of two exposure groups based on the arterial suturing pattern chosen by the operating surgeon, without protocol-driven randomization. Preoperative assessment follows national kidney transplantation guidelines and includes detailed history, physical examination, laboratory investigations, and multimodal imaging of donors and recipients. Intraoperative management is standardized regarding donor nephrectomy technique, transplant approach, vascular anastomosis sites, ureteroneocystostomy, ischemia time recording, and immunosuppressive regimen. Postoperative follow-up extends for at least three months, with serial clinical evaluations, renal function tests, Doppler ultrasound, and radiologic imaging when indicated to detect vascular complications and characterize graft function trajectories over time. The primary goal is to determine whether one suturing pattern is associated with more favorable ischemia metrics and hemodynamic parameters, thereby informing best practice for vascular anastomosis in living donor kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing living donor kidney transplantation at Assiut Kidney Transplantation Unit since November 2015

Exclusion Criteria:

* Patients undergoing end-to-end arterial suturing with internal iliac artery
* Patients with acute allograft rejection within the first post-transplant week
* Patients with follow-up shorter than 3 months after transplantation
* Patients with missing relevant preoperative or postoperative data
* Patients refusing participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study includes adult recipients of living donor kidney transplants performed at Assiut University Urology Hospital. Patients are selected based on having undergone or scheduled for living donor kidney transplantation, excluding those with end-to-end arterial suturing with the internal iliac artery, early acute rejection, or inadequate follow-up or data. Both retrospective cases and prospectively recruited patients with complete clinical, radiological, and laboratory data are included. The sample size is 70 patients divided equally between two arterial suturing technique groups.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Cold Ischemia Time | From donor graft perfusion to arterial de-clamping during the transplant operation (single intraoperative measurement).
  Duration in minutes from the start of graft perfusion with cold preservation solution in the donor to arterial de-clamping in the recipient, compared between interrupted and continuous arterial suturing groups.
Early Graft Arterial Blood Flow (Resistive Index and Systolic Velocity) | Within the first 3 months after transplantation (assessments at approximately 1 week, 1 month, and 3 months post-transplant).
  Mean systolic blood flow velocity and resistive index of the transplanted kidney artery measured by Doppler ultrasound and compared between interrupted and continuous arterial suturing groups.